CLINICAL TRIAL: NCT02306798
Title: An Open Label, Single-site Pharmaco-Scintigraphic Study in Healthy Subjects With Radio-labelled TP05-tablets (Mesalazine) to Evaluate the Gastrointestinal Transit and Release Profile
Brief Title: TP0502-B-Pharmaco-Scintigraphic-Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Tillotts Pharma AG (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: TP0502 - B
Record Dates: First submitted 2014-10-15; First posted 2014-12-03 (Estimated); Last update posted 2014-12-04 (Estimated); Status verified 2014-11

CONDITIONS: Ulcerative Colitis
MeSH Terms: conditions — Colitis, Ulcerative | interventions — Mesalamine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Formulation D (Experimental): TP05
  Interventions: Drug: TP05

INTERVENTIONS:
Drug: TP05 — One radio-labelled tablet given to subject after a high fat and a rich in calories breakfast
  Other Names: Mesalazine

SUMMARY:
This is a Phase I, open-label, single-site trial to evaluate the drug release, using scintigraphic images and mesalazine plasma levels (PK) in healthy subjects. Overall, nine [9] subjects will be evaluated. The subjects will receive one [1] radio-labelled tablet after a high fat and a rich in calories breakfast.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy subjects, male or non-pregnant, non-lactating females, between 18 and 55 years old. Females of child bearing potential must have a negative serum pregnancy test prior to the intake of study drug, and must use a hormonal (oral, implantable or injectable) or a double barrier method of birth control throughout the study. Females unable to bear children must have documentation of such in the source records (i.e., tubal ligation, hysterectomy, or post-menopausal [defined as a minimum of one year since the last menstrual period]).
2. Ability of subject to participate fully in all aspects of this clinical trial.
3. Written informed consent must be obtained and documented.

Exclusion Criteria:

1. Participating in a clinical study involving investigational drugs or dosage forms within the previous 30 days.
2. History of alcohol or drug abuse.
3. Radiation exposure from clinical trials, including that from the present study and from diagnostic X-ray but excluding background radiation, exceeds 5 mSv (milli-Sievert) in the last five years. No subject whose occupational exposure is monitored will participate in the study.
4. Any nuclear medicine procedure prior to study day 1 that might interfere with the scintigraphic images that are acquired.
5. Clinically significant abnormal biochemistry, haematology or urinalysis:

   * White blood count <3 x 109/L and >8 x 109/L
   * Lymphocyte count < 0.85 x 109/L
   * Haemoglobin < 110g/L
   * Platelet count < 125 x 109/L or > 600 x 109/L
   * Alanine-Aminotransferase (ALT) or Aspartate-Aminotransferase (AST) > 2x upper limit of normal
   * Alkaline Phosphatase > 2x upper limit of normal
   * Serum Creatinine > upper limit of normal
6. History of gastrointestinal surgery, with the exception of appendectomy unless it was performed within the previous 12 months.
7. History of cardiovascular, renal, hepatic, respiratory and particularly gastrointestinal disease, especially peptic ulceration, gastrointestinal bleeding, ulcerative colitis, Crohn's disease or Irritable Bowel Syndrome (within the previous 12 months).
8. Acute diarrhoea or constipation in the 14 days before the predicted first study day. If screening occurs >14 days before first study day, this criterion is to be determined on the first study day. Diarrhoea will be defined as the passage of liquid faeces and/or a stool frequency of greater than three times per day. Constipation will be defined as a failure to open the bowels more frequently than every other day.
9. History of adverse reaction or allergy to aspirin, mesalazine or other salicylates.
10. Donation of blood within the previous three months.
11. Positive HBV-Antigen (Hepatitis-B), HCV-Antibody (Hepatitis-C) or HIV-antibody (Human Immunodeficiency Virus) result.
12. Over-the-counter (OTC) and prescription medication (including laxatives, vitamins and natural herbal remedies) between screening visit (visit 1) and completion of the study. Occasional paracetamol or acetyl-salicylic acid is permitted.
13. Failure to satisfy the Principal Investigator to participate for any other reason.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 9 (Actual)
Dates: Start 2013-09; Primary Completion 2013-11 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Tablet release | 3 days

SECONDARY OUTCOMES:
Maximal Plasma Concentration (Cmax) | 3 days
Time to reach Cmax (Tmax) | 3 days
Area under the concentration time-curve | 3 days
Elimination rate konstant (k) | 3 days
Lag-time (t-lag) | 3 days